CLINICAL TRIAL: NCT04704180
Title: The Effect of Facilitated Tucking in the Early Postpartum Period on Preterm Neonatal Comfort and Breastfeeding Performance: A Randomized Controlled Trial
Brief Title: Facilitated Tucking Position's Effect on Comfort and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Assoch Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/319
Record Dates: First submitted 2021-01-02; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Breastfeeding, Exclusive; Position; Preterm Birth
Keywords: Facilitated tucking; breastfeeding performance; comfort; Preterm
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Intervention Model Description: In this study, stratified sampling was employed based on Gestational age. Two strata, [35-(35+6 days)] and [36-(36+6 days)], were generated to ensure even distribution in terms of Gestational age in each group. First, ninety-two preterm neonates were stratified into two groups (A and B), which were then stratified again into two: [35-(35+6 days)] and [36-(36+6 days)].
  A scheme was developed to randomize the gestational weeks of [35-(35+6 days)] and [36-(36+6 days)] into two groups (A and B), resulting in the experimental and control groups stratified by the week of gestation and blocked into paired-groups of (2:2/[35-(35+6 days)]:[36-(36+6 days)]). Permutation was also used to strike a balance between the strata. Block sets were generated for each combination of the prognostic factors (gestational age). The experimental and control groups were then randomized into the strata using a random numbers table.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Facilitation Tuchking Group (Experimental): The experimental group neonates received facilitated tucking under the radiant heater after birth of the NICU as well as the routine interventions.
  Interventions: Behavioral: Facilitation Tuchking Position
- Control Group (No Intervention): The control group underwent the routine interventions of the observation unit of the NICU. The group did not receive any other intervention

INTERVENTIONS:
Behavioral: Facilitation Tuchking Position — The nurse placed the neonate in the facilitated tucking position by rolling up a sizeable sterile towel in a U-shape and covering it with covers available in the unit and then placed the neonate in a supine position. The physiological parameters at admission and in the 15th and 30th minutes of facilitated tucking were recorded. In the 30th minute of facilitated tucking, the researcher and the observer nurse completed the COMFORTneo simultaneously but separately. The neonate was in the facilitated tucking position until delivered to its mother. The researcher and the observer nurse had a full view of the neonate's face and body when completing the COMFORTneo, which took them about two minutes. After the neonate stabilized (within the first half an hour to an hour), it was delivered to its mother for breastfeeding based on specialist consent. The first breastfeeding was performed and completed the LATCH by researcher and the observer nurse.
  Arms: Experimental Group: Facilitation Tuchking Group

SUMMARY:
This study investigated the effect of facilitated tucking in the early postpartum period on preterm neonate comfort and breastfeeding performance.

DETAILED DESCRIPTION:
Individualized Developmental Care (IDC) offered by NICUs yields positive outcomes in preterm neonates and neonates. Those positions should be comfortable and safe to promote physiological stability and optimal neuromotor development. The facilitated tucking position is the position of the baby in its mother's womb. It calms the neonate and helps it feel safe and maintain body control. It also improves sleep quality, stabilizes physiological parameters, gives a sense of security, supports motor development, and optimizes energy use. The facilitated tucking position makes it easier for preterm neonates to undergo invasive procedures (heel blood collection, aspiration etc.). However, there is no published research examining the effect of the facilitated tucking position in the early postpartum period on physiological parameters, comfort, and breastfeeding performance in preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* Born at 35-37 weeks of gestation,
* Appropriate weight for the week of gestation,
* 1-min and 5-min Apgar score of ≥ 8,
* No oxygen therapy,
* No anatomical and physiological problems,
* Showing no signs of illness,
* No congenital disorder,
* No breastfeeding problems

Exclusion Criteria:

* No parental consent
* Medical intervention other than the follow-up

Ages: 35 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Physiological Parameter Follow-up Form | First measurement- After admission in NICU 15th minutes
  The descriptive characteristics form was based on a literature review conducted by the researcher (Axelin, Salanterä & Lehtonen, 2006; Kucukoglu, Kurt & Aytekin, 2015; Yin, Yang, Lee, Li, Hua & Liaw, 2015). Heart rate (min), oxygen saturation (SpO2%), body temperature (°C), and respiration rate (min) was measured at admission to the NICU at 15th minutes
Physiological Parameter Follow-up Form | Secont measurement- After admission in NICU 30th minutes
  Heart rate (min), oxygen saturation (SpO2%), body temperature (°C), and respiration rate (min) was measured at admission to the NICU at 30th minutes.
COMFORT Behavior Scale for Neonates | In the 30th minute
  The COMFORT behavior scale for neonates (COMFORTneo) is a Likert-type measure of sedation and comfort needs, and pain and distress levels in NICU neonates. Van Dijk et al. (2009) established the validity and reliability of the COMFORTneo to measure only behavior in neonates. Kahraman, Başbakkal, and Yalaz (2014) adapted the scale to Turkish.
  In the 30th minute of facilitated tucking, the researcher and the observer nurse completed the COMFORTneo simultaneously but separately. The neonate was in the facilitated tucking position until delivered to its mother. The Intraclass Correlation Coefficient (ICC) was calculated to check the inter-observer agreement. The results indicated a perfect inter-observer agreement. The researcher and the observer nurse had a full view of the neonate's face and body when completing the COMFORTneo, which took them about two minutes.
LATCH | First breastfeeding (Within the first half an hour to an hour after birth).
  The LATCH breastfeeding diagnostic form was developed by Jensen, Wallace, and Kelsay (1994) and adapted to Turkish by Yenal and Okumuş (2003).
  Each letter of the acronym "LATCH" denotes a criterion for breastfeeding assessment: Latch onto the breast (L), audible swallowing (A), type of nipple (T), comfort (C), hold/help (H). The items are scored on a three-point Likert-type scale.
  After the neonate stabilized (within the first half an hour to an hour), it was delivered to the mother for breastfeeding based on specialist consent. The researcher and the observer simultaneously and independently observed the mother breastfeeding and completed the LATCH. The first breastfeeding was performed when the neonate was awake and active.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Principal Investigator — Selcuk Universty
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Result] Kahraman A, Basbakkal Z, Yalaz M, Sozmen EY. The effect of nesting positions on pain, stress and comfort during heel lance in premature infants. Pediatr Neonatol. 2018 Aug;59(4):352-359. doi: 10.1016/j.pedneo.2017.11.010. Epub 2017 Nov 13. PMID 29248383
- [Result] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525
- [Result] Axelin A, Salantera S, Lehtonen L. 'Facilitated tucking by parents' in pain management of preterm infants-a randomized crossover trial. Early Hum Dev. 2006 Apr;82(4):241-7. doi: 10.1016/j.earlhumdev.2005.09.012. Epub 2006 Jan 10. PMID 16410042
- [Result] Kucukoglu S, Kurt S, Aytekin A. The effect of the facilitated tucking position in reducing vaccination-induced pain in newborns. Ital J Pediatr. 2015 Aug 21;41:61. doi: 10.1186/s13052-015-0168-9. PMID 26293573
- [Result] Yin T, Yang L, Lee TY, Li CC, Hua YM, Liaw JJ. Development of atraumatic heel-stick procedures by combined treatment with non-nutritive sucking, oral sucrose, and facilitated tucking: a randomised, controlled trial. Int J Nurs Stud. 2015 Aug;52(8):1288-99. doi: 10.1016/j.ijnurstu.2015.04.012. Epub 2015 Apr 23. PMID 25939641
- [Derived] Altay G, Kucukoglu S. Effects of the facilitated tucking position in early period on physiological parameters, comfort and breastfeeding performance in late preterm infants: A randomized controlled trial. Midwifery. 2022 Dec;115:103492. doi: 10.1016/j.midw.2022.103492. Epub 2022 Sep 23. PMID 36201966